CLINICAL TRIAL: NCT00004800
Title: Phase III Randomized, Double-Blind, Placebo-Controlled Study of Acellular and Whole-Cell Pertussis Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Collaborators: Istituto Superiore di Sanità (Other)
Organization: Office of Rare Diseases (ORD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Prevention
Other Study IDs: 199/11954; ISS-RI-11954
Record Dates: First submitted 2000-02-24; First posted 2000-02-25 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-02

CONDITIONS: Pertussis
Keywords: bacterial infection; immunologic disorders and infectious disorders; pertussis; rare disease
MeSH Terms: conditions — Whooping Cough; Bacterial Infections; Immune System Diseases; Communicable Diseases; Rare Diseases | interventions — Diphtheria-Tetanus Vaccine

INTERVENTIONS:
Biological: diphtheria-tetanus-pertussis vaccine containing whole-cell pertussis
Biological: diphtheria-tetanus vaccine

SUMMARY:
OBJECTIVES: I. Compare the efficacy of 2 acellular pertussis vaccines vs. whole-cell pertussis vaccine vs. placebo in infants living in Italy.

II. Compare the relative protection of each of the acellular vaccines vs. the whole-cell vaccine vs. laboratory-confirmed pertussis.

III. Assess the relative efficacy of the acellular vaccines with respect to one another.

IV. Assess the immunogenicity of acellular vs. whole-cell vaccines in the study population.

V. Compare the frequency of adverse events with each vaccine. VI. Compare the frequency of adverse events attributable to the pertussis component in each of the 3 vaccines.

VII. Assess alternative laboratory diagnostic techniques for pertussis in estimating vaccine efficacy, i.e., mucosal immune response, DNA probes, or antibody response to other components of the organism.

VIII. Assess the relative efficacy estimates of each vaccine, using clinical criteria to compare the relative incidence rates in each vaccine group.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: This is a randomized, double-blind study. Patients are stratified by participating institution and randomly assigned to 1 of 3 vaccines and a placebo vaccine in a 3:3:3:1 ratio.

One group receives diphtheria-tetanus-pertussis (DPT) vaccine containing filamentous hemagglutinin (FHA), Pt-9K/129G, and 69 kDA outer membrane protein (OMP).

A second group receives DPT containing FHA and OMP. The third group receives DPT containing whole-cell pertussis. The control group receives diphtheria-tetanus (DT) vaccine. All vaccines are administered as an intramuscular or deep subcutaneous injection at 6-12, 13-20, and 21-28 weeks of age. The first vaccine is given at week 12 if hepatitis B or other immune globulin was given at birth.

All patients receive a DT booster at 11 months, and are followed every 4 weeks for approximately 20 months.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Population Characteristics-- Newborns enrolled at first vaccine clinic visit Weight at first vaccination at least third percentile, i.e.: Girls: 3.2 to 3.8 kg Boys: 3.4 to 4.0 kg No previous illness compatible with pertussis --Prior/Concurrent Therapy-- No prior pertussis vaccination --Patient Characteristics-- Age: Over 6 weeks to under 12 weeks Renal: No renal failure Other: No prior prolonged immunosuppressive therapy No prior systemic corticosteroids, unless duration less than 14 days and at least 48 hours since last dose No major congenital abnormality No failure to thrive No known or possible immune system deficit, e.g.: HIV-infected mother Autoimmune anemia Lymphoma Other erythropoietic disease No perinatal central nervous system disease or damage No history of convulsions Mother Italian-speaking and accessible by telephone Planned residence in clinic district for at least 1 year

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 13250
Dates: Start 1992-09

CONTACTS AND LOCATIONS:
Overall Officials: Donato Greco, Study Chair — Istituto Superiore di Sanità

REFERENCES:
- [Background] Greco D, Salmaso S, Mastrantonio P, Giuliano M, Tozzi AE, Anemona A, Ciofi degli Atti ML, Giammanco A, Panei P, Blackwelder WC, Klein DL, Wassilak SG. A controlled trial of two acellular vaccines and one whole-cell vaccine against pertussis. Progetto Pertosse Working Group. N Engl J Med. 1996 Feb 8;334(6):341-8. doi: 10.1056/NEJM199602083340601. PMID 8538704